CLINICAL TRIAL: NCT04542707
Title: Brainwave Activity Response on Common Physical Therapy Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida Gulf Coast University (Other)
Responsible Party: Principal Investigator, Dr. Rob Sillevis,, Assistant Professor, Florida Gulf Coast University
Allocation: Non-Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 2020-64
Record Dates: First submitted 2020-08-26; First posted 2020-09-09 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Pain
Keywords: Brain wave activity; Exercise; Joint manipulation; Soft tissue massage; Pupillometry
MeSH Terms: conditions — Pain; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: This experiment will be cross sectional study. Convenience sampling technique asymptomatic healthy subjects
Who Masked: Investigator, Outcomes Assessor
Masking Description: The treating clinician will not be aware off the brainwave and pupilometry data
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Joint manipulation (Experimental): Grade V-Thrust manipulation with audible sound and without audible sounds of C1-C2, T7, MTP 2 and MCP2 joints.
  Interventions: Procedure: joint manipulation
- Exercise (Experimental): Aerobic, anaerobic, and yoga exercises
  Interventions: Procedure: Exercise
- Soft tissue massage (Experimental): Instrument assisted soft tissue massage
  Interventions: Device: Soft tissue massage

INTERVENTIONS:
Procedure: joint manipulation — Thrust manipulation to the spine, hand, and foot
  Arms: Joint manipulation
Procedure: Exercise — Strength training, bike aerobic training, and yoga exercise
  Arms: Exercise
Device: Soft tissue massage — Graston tool
  Arms: Soft tissue massage

SUMMARY:
This study is designed to evaluate the if there is a predictable patterns in brainwave activity and to see how this changes with external physical therapy interventions such as manipulation, soft tissue massage, and exercise.

DETAILED DESCRIPTION:
This study is designed to evaluate the how the brain responds to external stimulation. Patients with chronic pain can benefit from physical therapy treatments, such as manipulation, soft tissue massage, and exercise. This study is made up of three different phases.

In the first phase to objective is to identify if there is a typical resting brain wave activity (measured with EEG) in asymptomatic subjects. In the second phase of the project the subjects will undergo physical therapy interventions and the brain wave response will be measured. The interventions are chosen based on the fact that they have been demonstrated in the literature to decrease pain.

Joint manipulation is a manual therapy intervention used with patients that experience pain and decreased range of motion. When undergoing a manipulation, audible sounds often occurring with the manipulation and sometimes this does not occur. In the current literature there is a difference between the effects of spinal manipulation and manipulation of the joints in the extremities. For that reason, this study will evaluate the response in both. It is not clear in the current literature if the audible sound has a true therapeutic effect. It is possible that patient perception of this sound will create a specific brainwave response pattern. This might support the clinician's pursuit of the audible sound.

Exercise has been shown to decrease pain, stiffness and increase ROM. Overall exercise contributes to wellbeing. There are different types of exercise such as strength exercise, aerobic exercise (aiming at increasing your heart rate) and body/ mind exercises (Yoga). In this phase of the study brainwave response on each of these types of exercises will be evaluated.

Soft tissue massage is a modality that has been shown to increase blood flow and decrease pain. This change in pain perception should lead to an altered brain wave activity.

As part of the phase the brain wave response on joint manipulation, exercise, and soft tissue massage on asymptomatic subjects will be measured and compared to each other. The hypothesis is that there will be a predictable pattern of brain response in each intervention.

The third phase of this study is to repeat the measures and intervention in subjects that experience pain. The hypothesis is that there is an altered brainwave response compared to the asymptomatic group. Additionally, in this phase the investigators will measure the brainwave response of FGCU college athletes who sprained their ankle within three days of the injury.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be between the ages of 18-60.
* The subjects for the manipulation group should have no history of thoracic spine pain in the last 6 months, no thoracic spine injuries within the past 6 months.
* The subjects for the exercise groups should be novice exercisers that do not workout often and can tolerate a 15 minute moderate intensity exercises.

Exclusion Criteria:

* A history of concussion, traumatic brain injury, stroke, or any known central nervous system disorder TBI, or brain damage.
* The specific exclusion criteria are for the manipulation group is osteopenia/osteoporosis or any other conditions or medications that would lead to skeletal compromise.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2020-08-20 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Brain wave activity | 1 hour
  EEG power in alpha, beta, delta, and gamma bands
Pupilometry | 5 minutes
  ANS response by measuring pupil diameter with automatic device

CONTACTS AND LOCATIONS:
Overall Officials: Rob Sillevis, Principal Investigator — FGCU
Locations (1):
- Florida Gulf Coast University, Fort Myers, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided
Not sure at his time